CLINICAL TRIAL: NCT04546399
Title: A Phase 2 Study of Blinatumomab (NSC# 765986) in Combination With Nivolumab (NSC # 748726), a Checkpoint Inhibitor of PD-1, in B-ALL Patients Aged >/= 1 to < 31 Years Old With First Relapse
Brief Title: A Study to Compare Blinatumomab Alone to Blinatumomab With Nivolumab in Patients Diagnosed With First Relapse B-Cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06813; NCI-2020-06813 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL1821 (Other: Children's Oncology Group); AALL1821 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome; Recurrent B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Down Syndrome; Burkitt Lymphoma | interventions — Radiotherapy, Conformal; Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; calaspargase pegol; Asparaginase; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Hydrocortisone; hydrocortisone hemisuccinate; Spinal Puncture; Mercaptopurine; azathiopurine; Methotrexate; merphos; Nivolumab; pegaspargase; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Arm G (dexamethasone, blinatumomab, nivolumab,MTX) DS patients (Experimental): Patients receive dexamethasone PO or IV on days 1 and 8 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28, nivolumab IV over 30 minutes on days 11 of cycle 1 and day 3 of cycle 2, and MTX IT (for patients with CNS1/2 at relapse only) or ITT on day 1 of cycle 1 only and days 15 and 36 (for patients with CNS 3 at relapse only) (day 1 IT therapy may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Cycles repeat every 37 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate; Biological: Nivolumab
- Group 1, Arm A (dexamethasone, blinatumomab, MTX) (Experimental): ARM A: Patients receive dexamethasone PO or IV on days 1 and 8 of cycle 1, blinatumomab via continuous IV infusion on days 1-28 of cycles 1-2, MTX IT, cytarabine IT, or ITT IT on days 1, 15, and 36 of cycle 1 (MTX, cytarabine, and ITT on day 1 may be omitted if intrathecal therapy was given < 7 days prior to the start of this cycle), and MTX IT, cytarabine IT, or ITT IT on days 15 and 36 of cycle 2. Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study. (CLOSED TO ACCRUAL 9/19/2024)
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate
- Group 1, Arm B (dexamethasone, blinatumomab, MTX) (Experimental): Patients receive dexamethasone, blinatumomab, and MTX, cytarabine, or ITT as in Arm A. Patients also receive nivolumab IV over 30 minutes on days 11 and 25 of cycle 1 and days 1 and 15 of cycle 2. Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study. (CLOSED TO ACCRUAL 9/19/2024)
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate; Biological: Nivolumab
- Group 2, Arm C (dexamethasone, blinatumomab, MTX) (Experimental): Patients receive dexamethasone PO or IV on day 1 of cycle 1, blinatumomab via continuous IV infusion on days 1-28 of cycles 1 and 2, and methotrexate IT on days 1 and 15 of cycles 1 and 2 (day 1 may be omitted from cycle 1 if intrathecal therapy is given < 7 days prior to the start of this cycle). Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study. (CLOSED TO ACCRUAL 9/19/2024)
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Dexamethasone; Procedure: Lumbar Puncture; Drug: Methotrexate
- Group 2, Arm D (dexamethasone, nivolumab, blinatumomab, MTX) (Experimental): Patients receive dexamethasone, blinatumomab, and MTX as in Arm C. Patients also receive nivolumab IV over 30 minutes on days 11 and 25 of cycle 1 and days 1 and 15 of cycle 2. Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study. (CLOSED TO ACCRUAL 9/19/2024)
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Dexamethasone; Procedure: Lumbar Puncture; Drug: Methotrexate; Biological: Nivolumab
- Group 3, Arm E (dexamethasone, blinatumomab, MTX) (Experimental): See Outline section
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Pegcrisantaspase; Drug: Vincristine Sulfate
- Group 3, Arm F (dexamethasone, blinatumomab, nivolumab) (Experimental): See Outline section
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Biological: Nivolumab; Drug: Pegaspargase; Drug: Pegcrisantaspase; Drug: Vincristine Sulfate
- Group 4 Arm I (Dexamethasone, blinatumomab, nivolumab) (Experimental): Patients receive dexamethasone PO or IV on day 1 and 8 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28, nivolumab IV, over 30 minutes on day 11 of cycle 1 and day 3 of cycle 2 and MTX IT on days 1 of cycle 1 only and days 15 and 36 ( for patients with CNS1/2 at relapse only) or ITT on day 1 of cycle 1 only and days 15 and 36 (for patients with CNS 3 at relapse only) (day 1 IT therapy may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Cycles repeat every 37 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate; Biological: Nivolumab
- Group 4, Arm H (dexamethasone blinatumomab) (Experimental): Patients receive dexamethasone PO or IV on day 1 and 8 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28 and MTX IT on days 1 of cycle 1 only and days 15 and 36 ( for patients with CNS1/2 at relapse only) or ITT on day 1 of cycle 1 only and days 15 and 36 (for patients with CNS 3 at relapse only) (day 1 IT therapy may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Cycles repeat every 37 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Dexamethasone; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
  Arms: Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab)
Procedure: Biospecimen Collection — Undergo blood, urine and cerebrospinal fluid collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
  Arms: Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab); Group 4 Arm I (Dexamethasone, blinatumomab, nivolumab)
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm G (dexamethasone, blinatumomab, nivolumab,MTX) DS patients; Group 1, Arm A (dexamethasone, blinatumomab, MTX); Group 1, Arm B (dexamethasone, blinatumomab, MTX); Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab); Group 4 Arm I (Dexamethasone, blinatumomab, nivolumab); Group 4, Arm H (dexamethasone blinatumomab)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Hydrocortisone Sodium Succinate — Given IT
  Other Names: (11beta)-21-(3-Carboxy-1-oxopropyl)-11,17-dihydroxypregn-4-ene-3,20-dione, Monosodium Salt; A-Hydrocort; Buccalsone; Corlan; Cortisol Sodium Succinate; Cortop; Efcortelan; Emergent-EZ; Flebocortid; Hidroc Clora; Hycorace; Hydro-Adreson; Hydrocort; Hydrocortisone 21-Sodium Succinate; Hydrocortisone Na Succinate; Kinogen; Nordicort; Nositrol; Sinsurrene; Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
  Arms: Arm G (dexamethasone, blinatumomab, nivolumab,MTX) DS patients; Group 1, Arm A (dexamethasone, blinatumomab, MTX); Group 1, Arm B (dexamethasone, blinatumomab, MTX); Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab); Group 4 Arm I (Dexamethasone, blinatumomab, nivolumab); Group 4, Arm H (dexamethasone blinatumomab)
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab)
Drug: Methotrexate — Given IT, PO, and IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm G (dexamethasone, blinatumomab, nivolumab,MTX) DS patients; Group 1, Arm B (dexamethasone, blinatumomab, MTX); Group 2, Arm D (dexamethasone, nivolumab, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab); Group 4 Arm I (Dexamethasone, blinatumomab, nivolumab)
Drug: Pegaspargase — Given IM or IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
  Arms: Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab)
Drug: Pegcrisantaspase — Given IM or IV
  Other Names: Asparec; JZP 416; JZP-416; JZP416; mPEG-R-crisantaspase; Pegylated Erwinia asparaginase; Pegylated Recombinant L-asparaginase Erwinia chrysanthemi
  Arms: Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab)
Drug: Vincristine Sulfate — Given IV push or via infusion
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Group 3, Arm E (dexamethasone, blinatumomab, MTX); Group 3, Arm F (dexamethasone, blinatumomab, nivolumab)

SUMMARY:
This phase II trial studies the effect of nivolumab in combination with blinatumomab compared to blinatumomab alone in treating patients with B-cell acute lymphoblastic leukemia (B-ALL) that has come back (relapsed). Down syndrome patients with relapsed B-ALL are included in this study. Blinatumomab is an antibody, which is a protein that identifies and targets specific molecules in the body. Blinatumomab searches for and attaches itself to the cancer cell. Once attached, an immune response occurs which may kill the cancer cell. Nivolumab is a medicine that may boost a patient's immune system. Giving nivolumab in combination with blinatumomab may cause the cancer to stop growing for a period of time, and for some patients, it may lessen the symptoms, such as pain, that are caused by the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare event free survival post reinduction (EFS PR) between blinatumomab vs. blinatumomab/nivolumab in Group 4 patients aged ≥ 1 to <31 years old with first relapse of CD19+ B ALL.

II. To compare EFS PR (EFS post-reinduction) between consolidation with blinatumomab vs. blinatumomab/nivolumab in Group 3 patients aged >= 1 to < 31 years old with first relapse of CD19+ B ALL.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of blinatumomab/nivolumab in patients aged >= 1 to < 31 years old with first relapse of CD19+ B ALL.

EXPLORATORY OBJECTIVES:

I. In Group 4 patients, compare EFS PR between blinatumomab monotherapy and blinatumomab/nivolumab arms as compared to similar patients treated on the predecessor trial AALL1331.

II. In Group 4 patients, compare toxicity as defined by grade 3 or greater adverse events during the first cycle of blinatumomab or blinatumomab/nivolumab.

III. In Group 4 patients, compare MRD negative second remission (Rem-2) rate after the first cycle of immunotherapy between blinatumomab monotherapy and blinatumomab/nivolumab arms.

IV. In patients with Down syndrome (DS) with first relapse of B-ALL, describe the safety, tolerability and efficacy (as defined by MRD negative second remission, Rem-2) after up to two cycles of blinatumomab/nivolumab.

V. With each Group, perform subset analyses of EFS and overall survival (OS) based on features including degree of marrow disease at relapse, age, sex, body mass index, cytogenetics, site(s) of relapse, percent peripheral blasts at relapse and absolute lymphocyte count at first relapse.

OUTLINE:

Patients >= 18 years old with marrow +/- extramedullary (EM) relapse of any duration after initial diagnosis, or patients < 18 years old with marrow +/- EM relapse < 24 months after initial diagnosis are assigned to Group 1. Patients < 18 years old with marrow +/- EM relapse >= 24 months from initial diagnosis, or all isolated extramedullary (IEM) relapses >= 1 to < 31 years old are assigned to Groups 2-3 re-induction. Patients with DS are assigned to Arm G. NOTE: Patients in Group 1 and DS patients with white blood cells (WBC) >= 30,000/uL, CNS 2/3 disease, or testicular disease must first receive 1 of 3 pre-immunotherapy treatments.

Starting with amendment 4C (9/19/2024), patients with DS are assigned to group 3 or 4. Patients < 18 years with bone marrow first relapse ≥ 36 months from initial diagnosis with MRD <0.1% after VXLD reinduction or with isolated CNS/testicular extramedullary relapse occurring ≥ 18 months from initial diagnosis with MRD <0.1% after VXLD reinduction are assigned to group 3. Patients who do not meet criteria for group 3 will be assigned to group 4. Patients with Down syndrome ≥ 1 to < 31 years of age with first bone marrow relapse of B ALL are assigned to arm G.

PRE-IMMUNOTHERAPY TREATMENT FOR PATIENTS WITH WBC >= 30,000/uL (CLOSED TO ACCRUAL 9/19/2024 EXCEPT FOR ARM G) : Patients receive methotrexate (MTX) intrathecally (IT) or cytarabine IT or intrathecal triple therapy (ITT) consisting of MTX, hydrocortisone sodium succinate, and cytarabine IT at the time of diagnostic lumbar puncture (LP) or on day 1 (if intrathecal therapy is given with relapse diagnostic LP < 7 days prior to the start of protocol therapy). Patients also receive dexamethasone intravenously (IV) or orally (PO) twice daily (BID) on days 1-5, vincristine sulfate via infusion or IV push over 1 minute on day 1. Patients with DS also receive leucovorin calcium PO or IV every 6 hours (q6h) for 2 doses on day 2 or at 24 and 30 hours after each IT administration. Patients should proceed to the next cycle when CNS 1 and no testicular disease is present, no sooner than Day 8 and no later than Day 15.

PRE-IMMUNOTHERAPY TREATMENT FOR CNS 2/3 DISEASE (CLOSED TO ACCRUAL 9/19/2024 EXCEPT FOR ARM G): Patients receive MTX IT or cytarabine IT twice weekly (Q2W) for 5-7 doses or Intrathecal Triple Therapy (ITT) IT Q2W for 3-4 doses until patient is CNS 1. Patients with DS also receive leucovorin calcium PO or IV q6h for 2 doses at 24 and 30 hours after each IT administration. Patients should proceed to the next cycle when CNS 1 and no testicular disease is present, no sooner than Day 15 and no later than Day 24.

PRE-IMMUNOTHERAPY TREATMENT FOR TESTICULAR DISEASE(CLOSED TO ACCRUAL 9/19/2024 EXCEPT FOR ARM G): Patients receive MTX IT, cytarabine IT, or ITT IT on days 1 and 15 (day 1 may be omitted if intrathecal therapy is given with relapse diagnostic LP < 7 days prior to the start of protocol therapy). Patients with DS also receive leucovorin calcium PO or IV q6h for 2 doses on days 2 and 16 or at 24 and 30 hours after each IT administration. Males with testicular disease at relapse undergo radiation once daily (QD) for a total of 12 fractions over 12 days. Patients should proceed to the next cycle when CNS 1 and no testicular disease is present, no sooner than Day 15 and no later than Day 22.

GROUP 1 (CLOSED TO ACCRUAL 9/19/2024): Patients are randomized to Arm A or Arm B.

ARM A: Patients receive dexamethasone PO or IV on days 1 and 8 of cycle 1, blinatumomab via continuous IV infusion on days 1-28 of cycles 1-2, MTX IT, cytarabine IT, or ITT IT on days 1, 15, and 36 of cycle 1 (MTX, cytarabine, and ITT on day 1 may be omitted if intrathecal therapy was given < 7 days prior to the start of this cycle), and MTX IT, cytarabine IT, or ITT IT on days 15 and 36 of cycle 2. Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2.

ARM B: Patients receive dexamethasone, blinatumomab, and MTX, cytarabine, or ITT as in Arm A. Patients also receive nivolumab IV over 30 minutes on days 11 and 25 of cycle 1 and days 1 and 15 of cycle 2. Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2.

GROUPS 2-4 VXLD REINDUCTION: Patients receive vincristine sulfate via infusion or IV push over 1 minute on days 1, 8, 15, and 22, dexamethasone PO or IV on days 1-14, doxorubicin hydrochloride IV over 1-15 minutes on day 1, MTX IT on days 1, 8, and 29 (day 1 IT may be omitted if intrathecal therapy is given with relapse diagnostic LP < 7 days prior to the start of this cycle) (days 8 and 29 for CNS 1 patients at relapse only), pegaspargase intramuscularly (IM) or IV over 1-2 hours on days 2 and 16 or calaspargase IV over 1-2 hours on day 2 (for patients ≤ 22 years), cytarabine IT on days 4 and 11 (CNS 2 patients at relapse only), then Q2W until 3 consecutive samples are clear of blasts, and ITT IT on days 8, 15, 22, and 29 (CNS 3 patients at relapse only). Treatment continues in the absence of disease progression or unacceptable toxicity.

GROUP 2 (CLOSED TO ACCRUAL 9/19/2024): The following patients are randomized to Arm C or Arm D: 1) >= 1 to < 31 years old, IEM relapse < 18 months from diagnosis, regardless of MRD after Re-Induction. 2) < 18 years old with marrow relapse >= 24 to < 36 months from diagnosis regardless of MRD after Re-Induction, 3) >= 1 to < 31 years old, IEM relapse >= 18 months, and MRD >= 0.1% after Re-Induction, 4) < 18 years old with marrow relapse >= 36 months, and MRD >= 0.1% after Re-Induction.

ARM C: Patients receive dexamethasone PO or IV on day 1 of cycle 1, blinatumomab via continuous IV infusion on days 1-28 of cycles 1 and 2, and MTX IT on days 1 and 15 of cycles 1 and 2 (day 1 may be omitted from cycle 1 if intrathecal MTX is given < 7 days prior to the start of cycle 1 ). Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2.

ARM D: Patients receive dexamethasone, blinatumomab, and MTX as in Arm C. Patients also receive nivolumab IV over 30 minutes on days 11 and 25 of cycle 1 and days 1 and 15 of cycle 2. Treatment repeats every 36 days for 2 cycles in the absence of disease progression or unacceptable toxicity. NOTE: Patients with MRD < 0.01% after cycle 1 may stop study treatment or may choose to continue to cycle 2. Patients with MRD >= 0.01% after cycle 1 proceed to cycle 2.

GROUP 3: Patients are randomized to Arm E or Arm F.

ARM E:

IMMUNOTHERAPY CYCLES 1-2: Patients receive dexamethasone PO or IV on day 1 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28, and MTX IT on days 1 and 15 (day 1 may be omitted from cycle 1 if intrathecal therapy is given < 7 days prior to the start of this cycle). Immunotherapy cycles 1-2 alternate with Consolidation cycles 1-2.

CONSOLIDATION: Patients receive dexamethasone PO or IV on days 1-5, methotrexate IV, over 24 hours, on days 8 and 22, methotrexate IT on days 8 and 22 (CNS 1/2 at relapse only) or ITT IT on days 8 and 22 (CNS 3 at relapse only).

INTENSIFICATION CYCLES 1-2: Patients receive dexamethasone PO on days 1-5, vincristine sulfate IV push over 1 minute or via infusion on day 1, mercaptopurine PO on days 1-42, methotrexate IV over 24 hours on days 8 and 22, cytarabine IV, over 3 hours on days 43 and 44, asparaginase erwinia recombinant IM or crisantaspase/asparaginase erwinia IM or IV over 1-2 hours on day 44, methotrexate IT on days 1 and 43 (CNS 1/2 at relapse only) or ITT IT on days 1 and 43 (CNS 3 at relapse only).

IMMUNOTHERAPY CYCLE 3: Patients receive blinatumomab IV via continuous infusion on days 1-28, and MTX IT on days 1 and 15 (CNS 1/2 at relapse only) or ITT IT on days 1 and 15 (CNS 3 at relapse only).

MAINTENANCE: Patients receive dexamethasone PO BID on days 1-5, 29-33, and 57-61, vincristine sulfate IV push over 1 minute or via infusion on days 1, 29, and 57, mercaptopurine PO on days 1-84, MTX IT on day 1 (CNS 1/2 patients at relapse only), ITT IT on day 1 (CNS 3 patients at relapse only), and MTX PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 12 weeks for 2 years from the start of Re-Induction therapy in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CHEMORADIATION (FOR CNS 3 PATIENTS ONLY): Beginning between the first and second cycles of maintenance therapy, patients receive dexamethasone PO BID on days 1-7 and 15-21, vincristine sulfate IV push over 1 minute or via infusion on days 1, 8, and 15, and pegaspargase IM or IV over 1-2 hours or calaspargase IV over 1-2 hours on day 1. Patients with CNS 3 and isolated CNS relapse undergo cranial radiation in the form of 3-dimensional (D)-conformal radiation therapy (CRT) over 5 days per week for a total of 10 treatments.

ARM F:

IMMUNOTHERAPY CYCLES 1-2: Patients receive dexamethasone PO or IV on day 1 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28, nivolumab IV over 30 minutes on days 11 of cycle 1 and on days 1 of cycles 2 and 3, and MTX IT on days 1 and 15 (CNS 1/2 patients at relapse only)(day 1 may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle) or , ITT IT on day 1 (CNS 3 patients at relapse only) (day 1 may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Immunotherapy cycles 1-2 alternate with Consolidation cycles 1-2.

CONSOLIDATION CYCLES 1-2: Patients receive dexamethasone PO on days 1-5, vincristine sulfate IV push over 1 minute or via infusion on day 1, methotrexate IV, over 24 hours, on days 8 and 22, methotrexate IT on days 8 and 22 (CNS 1/2 at relapse only) or ITT IT on days 8 and 22 (CNS 3 at relapse only).

INTENSIFICATION CYCLES 1-2: Patients receive dexamethasone PO on days 1-5, vincristine sulfate IV push over 1 minute or via infusion on day 1, mercaptopurine PO on days 1-42, methotrexate IV over 24 hours on days 8 and 22, cytarabine IV, over 3 hours on days 43 and 44, asparaginase erwinia recombinant IM or crisantaspase/asparaginase erwinia IM or IV over 1-2 hours on day 44, methotrexate IT on days 1 and 43 (CNS 1/2 at relapse only) or ITT IT on days 1 and 43 (CNS 3 at relapse only).

IMMUNOTHERAPY CYCLE 3: Patients receive blinatumomab IV via continuous infusion on days 1-28, nivolumab IV over 30 minutes on days 1 and 15 and MTX IT on days 1 and 15.

MAINTENANCE: Patients receive dexamethasone PO BID on days 1-5, 29-33, and 57-61, vincristine sulfate IV push over 1 minute or via infusion on days 1, 29, and 57, mercaptopurine PO on days 1-84, MTX IT on day 1 (CNS 1/2 patients at relapse only), ITT IT on day 1 (CNS 3 patients at relapse only), and MTX PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78. Treatment repeats every 12 weeks for 2 years from the start of Re-Induction therapy in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CHEMORADIATION (FOR CNS 3 PATIENTS): Beginning between the first and second cycles of maintenance therapy, patients receive dexamethasone PO BID on days 1-7 and 15-21, vincristine sulfate IV push over 1 minute or via infusion on days 1, 8, and 15, and pegaspargase IM or IV over 1-2 hours or calaspargase IV over 1-2 hours on day 1. Patients with CNS 3 and isolated CNS relapse undergo cranial radiation in the form of 3-dimensional (D)-conformal radiation therapy (CRT) over 5 days per week for a total of 10 treatments.

GROUP 4: Patients are randomized to arm H or arm I.

ARM H: Patients receive dexamethasone PO or IV on day 1 and 8 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28 and MTX IT on days 1 of cycle 1 only and days 15 and 36 ( for patients with CNS1/2 at relapse only) or ITT on day 1 of cycle 1 only and days 15 and 36 (for patients with CNS 3 at relapse only) (day 1 IT therapy may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Cycles repeat every 36 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

ARM I: Patients receive dexamethasone PO or IV on day 1 and 8 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28, nivolumab IV, over 30 minutes on day 11 of cycle 1 and day 3 of cycle 2 and MTX IT on days 1 of cycle 1 only and days 15 and 36 ( for patients with CNS 1/2 at relapse only) or ITT on day 1 of cycle 1 only and days 15 and 36 (for patients with CNS 3 at relapse only) (day 1 IT therapy may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Cycles repeat every 36 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

ARM G (DS PATIENTS): Patients receive dexamethasone PO or IV on days 1 and 8 of cycle 1 only, blinatumomab IV via continuous infusion on days 1-28, nivolumab IV over 30 minutes on days 11 of cycle 1 and day 3 of cycle 2, and MTX IT (for patients with CNS 1/2 at relapse only) or ITT on day 1 of cycle 1 only and days 15 and 36 (for patients with CNS 3 at relapse only) (day 1 IT therapy may be omitted from cycle 1 if intrathecal therapy is given with < 7 days prior to the start of this cycle). Cycles repeat every 37 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo lumbar puncture, bone marrow biopsy and aspiration, and collection of blood, urine and cerebrospinal fluid throughout the study.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 1 and < 31 years at time of enrollment
* Patients must have first relapse of CD19+ B-ALL (relapse blasts must express CD19) in one of the following categories:

  * Isolated bone marrow relapse
  * Isolated central nervous system (CNS) (excluding known optic nerve/retinal and CNS chloromas) and/or testicular relapse
  * Combined bone marrow with extramedullary relapse in the CNS (excluding known optic nerve/retinal and CNS chloromas) and/or testes
* Patients with Down syndrome (DS) are eligible in the following categories:

  * Isolated bone marrow relapse
  * Combined bone marrow with CNS (excluding known optic nerve/retinal and CNS chloromas) and/or testicular relapse
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age

  * Of note, for patients with developmental delay (e.g., Down syndrome) regardless of age, Lansky scale may be substituted for Karnofsky scale. However, the requirement for ECOG 0-2 remains, regardless of known history of developmental delay
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Patients with prior blinatumomab or CD19+ chimeric antigen receptor therapy in the upfront setting will be eligible, provided relapsed lymphoblasts retain CD19 expression
  * Patients must not have had a prior hematopoietic stem cell transplant
  * A single intrathecal chemotherapy at the time of relapse will be allowed. If < 7 days have elapsed between this intrathecal therapy (IT) and the start of protocol therapy, then the day 1 intrathecal chemotherapy (i.e. methotrexate, cytarabine, or triple intrathecal) may be omitted
  * In the 28 days prior to enrollment, up to five days of post-relapse, pre-enrollment therapy (steroids and/or hydroxyurea only) is permissible

    * Patients with Down syndrome who received pre-enrollment therapy and have a white blood count (WBC) >= 30,000/ul at the time of enrollment still must receive protocol specified cytoreductive therapy with vincristine and dexamethasone, and no "washout" is required
    * Patients with Down syndrome who received pre-enrollment therapy and have a WBC < 30,000/ul at the time of enrollment must be given a 24 hour "washout" before starting immunotherapy
  * Note: There is no waiting period or "washout" for patients who relapse while receiving upfront therapy
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/sex as follows (within 7 calendar days prior to enrollment):

  * Age: Maximum serum creatinine (mg/dL)

    * 1 to < 2 years: 0.6 (male), 0.6 (female)
    * 2 to < 6 years: 0.8 (male), 0.8 (female)
    * 6 to < 10 years: 1 (male), 1 (female)
    * 10 to < 13 years: 1.2 (male), 1.2 (female)
    * 13 to < 16 years: 1.5 (male), 1.4 (female)
    * >= 16 years: 1.7 (male), 1.4 (female)

      * The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Center for Disease Control (CDC)
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by echocardiogram, cardiac magnetic resonance imaging (MRI) or radionuclide angiogram
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with B-lymphoblastic lymphoma (B-LLy)
* Patients with Burkitt leukemia/lymphoma or mature B-cell leukemia
* Patients with Philadelphia chromosome positive (Ph+) B-ALL
* Patients with mixed phenotype acute leukemia (MPAL)
* Patients with known Charcot-Marie-Tooth disease
* Patients with known MYC translocation associated with mature (Burkitt) B-cell ALL, regardless of blast immunophenotype
* Patients with active, uncontrolled infection defined as:

  * Positive bacterial blood culture within 48 hours of study enrollment
  * Receiving IV or PO antibiotics for an infection with continued signs or symptoms. Note: Patients may be receiving IV or oral antibiotics to complete a course of therapy for a prior documented infection if cultures have been negative for at least 48 hours and signs or symptoms of active infection have resolved. For patients with clostridium (C.) difficile diarrhea, at least 72 hours of antibacterial therapy must have elapsed and stools must have normalized to baseline.
  * Fever above 38.2 degrees Celsius (C) within 48 hours of study enrollment with clinical signs of infection. Fever without clinical signs of infection that is attributed to tumor burden is allowed if blood cultures are negative for > 48 hours
  * A positive fungal culture within 30 days of study enrollment or active therapy for presumed invasive fungal infection
  * Active viral or protozoal infection requiring IV treatment
* Patients known to have one of the following concomitant genetic syndromes: Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome are not eligible.
* Patients with uncontrolled HIV, hepatitis B, or hepatitis C infection. Of note, patients with known human immunodeficiency virus (HIV) infection on effective anti-retroviral therapy with undetectable viral load for at least the last 6 months prior to enrollment are eligible. Similarly, hepatitis B and hepatitis C positive patients who have been treated and have no viral detectable burden are also eligible
* Patients with significant central nervous system pathology that would preclude treatment with blinatumomab, including history of severe neurologic disorder or autoimmune disease with CNS involvement

  * Note: Patients with a history of seizures that are well controlled on stable doses of anti-epileptic drugs are eligible Patients with a history of cerebrovascular ischemia/hemorrhage with residual deficits are not eligible. Patients with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits have resolved
* Patients with an active known/suspected autoimmune disease are not eligible. However, patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Group 4 and patients with DS patients with known non-hematopoietic, non-CNS/testicular extramedullary disease (i.e., chloromatous disease) are not eligible

  * Note: Group 3 patients with known non-hematopoietic, non-CNS/testicular extramedullary disease (i.e., chloromatous disease) are eligible if this is NOT the only site of relapsed disease
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained within 7 days prior to enrollment. Patients who are sexually active and of reproductive potential are not eligible unless they agree to use an effective contraceptive method for the duration of this study. Men with female partners of childbearing potential should use effective contraception during the duration of their treatment. The effect of blinatumomab on fertility has not been evaluated. Blinatumomab is not recommended for pregnant women or women of childbearing potential (WOCBP) not using contraception. Females of reproductive potential must use effective contraception during treatment and for at least 48 hours after the last dose of blinatumomab. Studies in animal models have shown that nivolumab can adversely impair pregnancy. Thus, nivolumab is expected to cause fetal harm during pregnancy. WOCBP receiving nivolumab must continue contraception for a period of at least 5 months after the last dose of nivolumab. It is unknown whether nivolumab is present in breast milk, thus breastfeeding should be discontinued while a patient is receiving nivolumab
* Lactating females are not eligible unless they agree to not breastfeed their infants. It is unknown whether blinatumomab or its metabolites are excreted in human breast milk. Women are not permitted to breastfeed while receiving blinatumomab and for the last 48 hours after the last blinatumomab dose. Due to the potential for serious adverse reactions in the breastfed infant, women are not permitted to breastfeed during treatment and for 5 months after the last nivolumab dose

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 461 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negative second remission (Rem-2) rate with blinatumomab vs with blinatumomab + nivolumab (Group 1) | Up to 2 cycles of therapy (each cycle = 36 days)
  MRD negative Rem-2 be defined as Rem-2 (i.e., achievement of MRD < 1% blasts by flow cytometry and resolution of extramedullary disease (for CNS disease, requires CNS 1) ) and bone marrow with MRD < 0.01% by flow cytometry. MRD negative Rem-2 rate between Arm A vs Arm B will be compared using a one-sided Z test of proportions with Type I error of 0.10. Interim analysis will be conducted to monitor for futility. The futility boundaries are based on testing the alternative hypothesis at the 0.067 level.
Event-free survival post-reinduction (EFS PR) (Group 3) | From date of randomization to date of treatment failure, relapse, disease progression, second malignancy (SMN) or death due to any cause, assessed up to 10 years after completion of enrollment.
  Comparison of EFS post reinduction between Arm E versus Arm F will be based on a one-sided two-sample logrank test with Type I error of 0.10, to be conducted 3 years after completion of enrollment of Group 3. Interim analysis will be conducted to monitor for futility. The futility monitoring will be based on testing the alternative hypothesis at the 0.067 level. This alpha level corresponds to that which would cause futility stopping if the one-sided two-sample logrank test shows evidence of a hazard ratio > 1.0 when half of the expected events are observed.
EFS PR (Group 4) | From date of randomization to date of treatment failure, relapse, disease progression, second malignancy (SMN) or death due to any cause, assessed up to 10 years after completion of enrollment.
  Comparison of EFS post reinduction between Arm H versus Arm I will be based on a one-sided two-sample logrank test with Type I error of 0.10, to be conducted 3 years after completion of enrollment of Group 3. Interim analysis will be conducted to monitor for futility. The futility monitoring will be based on testing the alternative hypothesis at the 0.067 level. This alpha level corresponds to that which would cause futility stopping if the one-sided two-sample logrank test shows evidence of a hazard ratio > 1.0 when half of the expected events are observed.

SECONDARY OUTCOMES:
Dose-limiting toxicity | Up to 1 cycle of therapy (each cycle = 36 days)
  Will be assessed using the Common Terminology Criteria for Adverse Events version 5.0.
EFS PR (Group 4) | From date of randomization to date of treatment failure, relapse, disease progression, SMN or death due to any cause, assessed up to 5 years after completion of enrollment
  Comparison of EFS post-reinduction between Arm C versus Arm D will be based on a one-sided two-sample logrank test with type I error of 0.15, to be conducted 2 years after completion of enrollment of Group 2. The futility monitoring will be based on testing the alternative hypothesis at the 0.092 level.

OTHER OUTCOMES:
Event-free survival (Group 1) | From date of Group 1 randomization to date of treatment failure, relapse, disease progression, SMN or death due to any cause, assessed up to 5 years
  EFS will be compared between Arm A and Arm B, and to similar patients treated on AALL1331. These analyses will be performed using logrank tests, semi-parametric or parametric survival analysis methods, as appropriate.
Event free survival (Group 4) | From date of Group 4 randomization to date of treatment failure, relapse, disease progression, SMN or death due to any cause, assessed up to 5 years
  EFS will be compared between Arm H and Arm I, and to similar patients treated on AALL1331. These analyses will be performed using logrank tests, semi-parametric or parametric survival analysis methods, as appropriate.
Incidence of adverse events in Arm A or Arm B | Up to 1 cycle of therapy (each cycle = 36 days)
  The toxicities as defined by grade 3 or greater reported adverse events during the first cycle of blinatumomab or blinatumomab/nivolumab will be compared to similar patients treated with Block 1 of cytotoxic chemotherapy on AALL1331 using two-sample test of proportions.
Incidence of adverse events in Arm H or Arm I | Up to 1 cycle of therapy (each cycle = 36 days)
  The toxicities as defined by grade 3 or greater reported adverse events during the first cycle of blinatumomab or blinatumomab/nivolumab will be compared to similar patients treated with Block 1 of cytotoxic chemotherapy on AALL1331 using two-sample test of proportions.
MRD negative Rem-2 rate (Group 2) | Up to 2 cycles of therapy (each cycle = 36 days)
  MRD negative Rem-2 rate will be estimated and be compared between Arm C and Arm D using two-sample test of proportions.
Dose-limiting toxicity (Down syndrome patients) | Up to 1 cycle of therapy (each cycle = 36 days)
  Analyses will be largely descriptive.
Incidence of adverse events (Down syndrome patients) | Up to 1 cycle of therapy (each cycle = 36 days)
  Analyses will be largely descriptive.
MRD negative Rem-2 rate (Down syndrome patients) | Up to 2 cycles of therapy (each cycle = 36 days)
  Analyses will be largely descriptive.
Subset analyses of EFS | Up to 2 cycles of therapy (each cycle = 36 days)
  Features at first relapse including degree of marrow disease at relapse, age, sex, body mass index, cytogenetics, site(s) of relapse, percent peripheral blasts at relapse and absolute lymphocyte count, will be conducted. These analyses will be exploratory.
Subset analyses of OS | Up to 2 cycles of therapy (each cycle = 36 days)
  Features at first relapse including degree of marrow disease at relapse, age, sex, body mass index, cytogenetics, site(s) of relapse, percent peripheral blasts at relapse and absolute lymphocyte count, will be conducted. These analyses will be exploratory.
EFS PR (Group 4) | At 2 years from date of randomization
  Corresponding 95% CIs by sex, by race, and by ethnicity separately for arm H and I.
EFS PR (Group 3) | At 3 years from date of randomization
  Corresponding 95% CIs by sex, by race, and by ethnicity separately for arm E and F.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy L Cooper, Principal Investigator — Children's Oncology Group
Locations (215):
- United States (202):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (7):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074